CLINICAL TRIAL: NCT06898463
Title: Comparison Of The Effects Of Melatonin Premedication And Ketamine On Postoperative Sleep Quality İn Rhinoplasty: A Prospective Randomized Controlled Study
Brief Title: Comparison Of The Effects Of Melatonin Premedication And Ketamine On Postoperative Sleep Quality İn Rhinoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konya City Hospital (Other)
Collaborators: necmettin erbakan university Scientific Research Projects (BAP) (Unknown)
Responsible Party: Principal Investigator, Ömer Keklicek, Principal Investigator MD, Konya City Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2022/927
Record Dates: First submitted 2025-03-12; First posted 2025-03-27 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Sleep Disturbances
Keywords: Rhinoplasty; Sleep Disorder; Melatonin; Ketamine
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Melatonin; Ketamine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- M GROUP (Active Comparator): In Group 1 (Melatonin, M), patients received 0.1 mg/kg oral melatonin 60 minutes before surgery in the premedication room and at 9 PM on the first postoperative day.
  Interventions: Drug: Melatonin (N-acetyl-5-methoxytryptamine)
- K GROUP (Active Comparator): In Group 2 (Ketamine, K), patients were administered 0.3 mg/kg intravenous ketamine during anesthesia induction.
  Interventions: Drug: Ketamine
- M-K GROUP (Active Comparator): In Group 3 (Melatonin-Ketamine, MK), patients received 0.1 mg/kg oral melatonin in the premedication room 60 minutes before surgery and at 9:00 PM on the first postoperative day, and 0.3 mg/kg intravenous ketamine during anesthesia induction.
  Interventions: Drug: Melatonin (N-acetyl-5-methoxytryptamine); Drug: Ketamine

INTERVENTIONS:
Drug: Melatonin (N-acetyl-5-methoxytryptamine) — 0.1 mg/kg oral melatonin was administered twice
  Arms: M GROUP; M-K GROUP
Drug: Ketamine — 0.3 mg/kg intravenous ketamine was administered during anesthesia induction.
  Arms: K GROUP; M-K GROUP

SUMMARY:
Background Postoperative sleep disorders are common complications of surgery and anesthesia that prolong morbidity and hospital stay. Various methods are being explored to prevent and treat these issues. This study was designed to investigate the effects of ketamine, melatonin, and their combination on postoperative sleep disturbances and pain.

Methods Patients were randomly allocated into three groups: melatonin (Group M), ketamine (Group K), and a melatonin-ketamine combination (Group MK). Group M received 0.1 mg/kg oral melatonin preoperatively (60 minutes before surgery) and postoperatively at 21:00; Group K received 0.3 mg/kg IV ketamine during anesthesia induction; and Group MK received both regimens. Sleep quality was assessed on the first postoperative day using the Richards-Campbell Sleep Questionnaire (RCSQ), and pain intensity was evaluated with the Numeric Rating Scale (NRS). Early extubation-related complications (e.g., coughing, breath-holding, desaturation, vomiting, and laryngospasm) and delayed complications in the post-anesthesia care unit (PACU) were documented. Demographic variables, including ASA physical status scores, were recorded. Intraoperative monitoring comprised basal, post-intubation, and post-extubation measurements of heart rate (HR), systolic arterial pressure (SAP), diastolic arterial pressure (DAP), and mean arterial pressure (MAP) at 30-minute intervals, together with recording surgery and extubation durations.

DETAILED DESCRIPTION:
Participants Patients aged 18-65 years with an ASA score of I-II were included. Exclusion criteria were body mass index (BMI) ≥ 30 kg/m², obstructive sleep apnea syndrome (OSAS), psychiatric disorders, renal failure, liver failure, cardiovascular disease, malignancy, pregnancy, or allergies to melatonin or ketamine. Randomization (1:1:1) was achieved via sealed opaque envelopes.

Interventions Patients were premedicated in the preoperative holding area 60 minutes before induction with intravenous midazolam (0.01 mg/kg), and subjects in Groups M and MK additionally received oral melatonin (0.1 mg/kg). After premedication, each patient was transferred to the operating theater, where continuous electrocardiography, pulse oximetry, noninvasive arterial pressure monitoring, and neuromuscular transmission (NMT) monitoring were applied. Anesthesia was induced with intravenous propofol (2 mg/kg), lidocaine (1 mg/kg), and rocuronium (0.6 mg/kg); at this point, patients in Groups K and MK received a supplemental ketamine bolus (0.3 mg/kg). Following confirmation of full neuromuscular blockade (train-of-four ratio = 0 %) and adequate hypnotic depth, endotracheal intubation was performed. Anesthesia was maintained with sevoflurane (0.5-1.0 minimum alveolar concentration [MAC] at a fresh gas flow of 1 L/min) and a remifentanil infusion (0.1-0.3 µg/kg/min). Dosages were titrated to maintain heart rate and systolic arterial pressure within 20-30 % of baseline values, ensuring mean arterial pressure did not fall below 50 mmHg.

Hemodynamic variables-including heart rate, systolic and diastolic arterial pressures, and mean arterial pressure-were recorded at four predefined time points: baseline (pre-induction), immediately post-intubation, at 30-minute intervals intraoperatively, and post-extubation. Thirty minutes before the end of surgery, postoperative analgesia was initiated with tramadol (2 mg/kg) and paracetamol (10 mg/kg) administered as slow intravenous boluses; ondansetron (0.1 mg/kg IV) was given prophylactically for nausea. Neuromuscular blockade was reversed, if necessary, with sugammadex to achieve a train-of-four ratio ≥ 90 %, and patients were extubated once adequate spontaneous ventilation and consciousness had returned. The extubation interval (time from anesthetic discontinuation to return of consciousness) and total surgical duration were documented. In the post-anesthesia care unit (PACU), nausea, vomiting, and pain scores were assessed; patients with moderate to severe nausea or vomiting received an additional 0.1 mg/kg ondansetron IV, and those reporting a resting numerical rating scale (NRS) pain score > 4 were given meperidine (0.5 mg/kg IV) as rescue analgesia. Finally, at 21:00 on postoperative day 1, Groups M and MK received a second oral dose of melatonin (0.1 mg/kg), and sleep quality and pain were re-evaluated at the bedside.

Outcomes Sleep quality was evaluated on the night preceding surgery and on the first postoperative night using the Richards-Campbell Sleep Questionnaire (RCSQ), which exhibits high internal consistency (Cronbach's α = 0.82) and correlates moderately with polysomnography. The RCSQ comprises five domains-sleep depth, sleep latency, number of awakenings, sleep efficiency, and overall sleep quality-each rated on a 0-100 mm visual analog scale, with higher scores indicating better sleep. Postoperative pain intensity was measured in the post-anesthesia care unit (PACU) and at 24 hours after surgery using an 11-point Numeric Rating Scale (NRS; 0 = no pain, 10 = worst imaginable pain).

Postoperative complications were recorded prospectively as follows: cough severity was graded by the Cough Severity Score (0 = none; 1 = mild; 2 = moderate; 3 = severe; 4 = very severe); apnea was defined as absence of a respiratory waveform for ≥ 10 seconds on capnography; desaturation was identified when SpO₂ fell below 90 % on continuous pulse oximetry; laryngospasm was classified according to the Laryngospasm Severity Scale (grade 1 = mild retraction; grade 2 = intercostal retractions; grade 3 = complete airway obstruction); and vomiting was quantified using the Rhodes Index of Nausea, Vomiting, and Retching (INVR). Finally, the Aldrete score was documented immediately before PACU discharge, and the interval from PACU admission to attainment of the discharge criterion was recorded.

Statistical Analysis Statistical analyses were performed using IBM SPSS Statistics v23.0 (IBM Corp., Armonk, NY, USA). Categorical variables are reported as frequencies and percentages and were compared by Pearson's chi-square or Fisher's exact test, as appropriate. Continuous variables were first assessed for normality using the Shapiro-Wilk test. Variables conforming to a normal distribution are presented as mean ± standard deviation and compared by one-way analysis of variance (ANOVA); homogeneity of variances was verified with Levene's test, and post hoc pairwise comparisons were conducted using Tukey's honestly significant difference or Games-Howell tests, as dictated by variance equality. Non-normally distributed variables are expressed as median (interquartile range) and were analyzed via the Kruskal-Wallis H test followed by Dunn's multiple-comparison test with Bonferroni adjustment. Sample size estimation using G*Power 3.1 (α = 0.05; 1 - β = 0.85; effect size f = 0.25) indicated that 60 patients per group were required. To allow for an anticipated 10% attrition rate, 200 patients were recruited; 17 were subsequently excluded (did not meet inclusion criteria or declined to participate), yielding a final sample of 183 participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients capable of providing consent
* Patients able to reliably report their symptoms to the research team
* Patients with American Society of Anesthesiologists (ASA) physical status I-II
* Patients aged 18-65 years
* Patients undergoing rhinoplasty surgery
* Exclusion Criteria:
* Patients with cognitive impairment or a communication barrier
* Patients with a BMI > 30
* Patients with OSAS (Obstructive Sleep Apnea Syndrome)
* Patients with a known psychiatric disorder
* Patients with renal failure
* Patients with liver failure
* Patients with cardiovascular disease (e.g., heart failure, coronary artery disease, arrhythmia, etc.)
* Patients with malignancy
* Patients who are pregnant or lactating
* Patients with a history of allergy to melatonin and ketamine
* Patients with an American Society of Anesthesiologists (ASA) Physical Status score ≥3
* Patients who do not consent to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
To compare the effects of melatonin and ketamine on postoperative sleep disturbances. | From enrollment to the end of treatment at 21 Mounths
  On postoperative day 1, patients' sleep quality was assessed at bedside using the Richards-Campbell Sleep Questionnaire (RCSQ). Although primarily used in intensive care settings, the RCSQ is also valid for assessing sleep in postoperative patients. It shows high internal consistency and moderate correlation with polysomnography. The RCSQ includes five items: sleep depth, latency, awakenings, efficiency, and overall quality. Each item is rated on a 0-100 mm visual analog scale, where higher scores reflect better sleep. The total score is the average of the five items.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University Faculty of Medicine, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Share the abstract and materials and methods section
Supporting Information: Study Protocol
Time Frame: starting in March 2025